CLINICAL TRIAL: NCT07037030
Title: The Investigation of a Mindfulness-Based Intervention for ADHD
Brief Title: Mindfulness ADHD Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, James Lynch, Postdoctoral Psychology Fellow, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00051676
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Breathing Intervention (Experimental): Children will complete a brief deep breathing intervention
  Interventions: Behavioral: Guided deep breathing

INTERVENTIONS:
Behavioral: Guided deep breathing — Children will complete a brief, 5-minute, deep breathing intervention using the Domi tool to help maintain a 5-second breath pace

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) affects approximately 11% of children and adolescents in the United States. Individuals with ADHD experience substantial impairments and burdens across multiple areas of daily living, including peer difficulties, academic difficulties, poor job outcomes, high rates of co-occurring disorders, and large financial costs. Although there are many well-established, evidence-based treatments for ADHD, many children continue to experience significant impairment and elevated ADHD symptoms even with prolonged treatment. Further, there are several limitations to existing treatment approaches, including medication side effects, difficulty accessing behavioral treatments, and high out-of-pocket costs for behavioral treatments. Thus, there is a crucial need to identify low cost, low burden, alternative or additive intervention approaches for pediatric ADHD.

In the current pilot study, we aim to evaluate responses in behavioral and brain-based markers of attention to a mindfulness-based intervention. Mindfulness-based interventions (MBIs), including deep breathing, have received considerable research attention regarding their benefits for ADHD symptoms. Deep breathing is a strong candidate as a supplementary MBI intervention for children with ADHD due to its simplistic and easy-to-implement nature. Studies examining the effects of deep breathing on physiological arousal and ADHD symptoms in children have yielded promising results. Children will be led through a brief deep breathing intervention using a novel tool designed to optimize child engagement in deep breathing. This tool, Domi, is designed to be held in the child's hands and uses a series of haptic vibrations to provide real-time deep breathing pacing guidance. We predict that following a brief deep breathing practice, children with ADHD will demonstrate improved sustained attention, reaction time consistency, and inhibitory control. These areas of attention and behavioral functioning will be assessed using computer tasks and measures of brain activity.

We plan to use the results of this study to strengthen a future application for grant funding to run a similar trial with many more children. We believe that the results of this and future studies will improve the lives of children with ADHD and their families.

ELIGIBILITY:
Inclusion Criteria:

* Participant age 7 years, 0 months - 11 years, 11 months
* Parent-reported ADHD diagnosis for the participant

Exclusion Criteria:

* Previous confirmed or suspected diagnosis of intellectual disability
* Previous confirmed or suspected diagnosis of autism spectrum disorder
* Currently prescribed non-stimulant medication for the purpose of managing ADHD symptoms
* Hearing impairments
* Primary language other than English
* Known seizure disorder

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Behavioral Performance Metrics | During the single in-person research visit
  Behavioral markers of sustained attention and inhibitory control will be assessed using a Go/NoGo task. Omission errors (failing to respond to a Go trial) and reaction time variability (standard deviation of reaction time across all trials) will serve as markers of sustained attention. Commission errors (responding to a NoGo trial) will serve as a marker of inhibitory control.
Neurophysiological Markers | During the single in-person research visit
  Electroencephalography (EEG) methods will be used to measure P300 event-related potentials (ERP), a positive inflection occurring around 300ms after a response to task-relevant and irrelevant stimuli that reflects attention orienting, stimulus evaluation, and inhibitory control. Stimulus-locked P300 amplitude in response to correct Go-trials will be a marker of cortical attention processes, while stimulus-locked P300 amplitude in response to NoGo trials will be a marker of cortical inhibitory control processes.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital Laboratories of Cognitive Neuroscience, Brookline, Massachusetts, United States